CLINICAL TRIAL: NCT00602966
Title: Oocyte Cryopreservation: Comparison of Slow Cooling Versus Vitrification Techniques on Oocyte Survival, Fertilization, and Embryo Development
Brief Title: Oocyte Cryopreservation: Slow Cooling Versus Vitrification Techniques on Oocyte Survival
Status: Completed | Type: Observational
Sponsor: UConn Health (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Principal Investigator, Claudio Benadiva, Laboratory Director and Director of the Preimplantation Genetics Diagnosis Program,, UConn Health
Other Study IDs: 06-336-2; 26525
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Infertility
Keywords: Oocyte cryopreservation; slow freeze; vitrification
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Slow Freeze
- Vitrification

SUMMARY:
Oocyte cryopreservation has been studied for many years without much success in refining a method that has consistent, reliable results in producing viable embryos and clinical pregnancies. In 1986 the first baby was born from an embryo created from a frozen oocyte; however, since then there have been less than 150 births from frozen eggs. To date, there are no reportable adverse outcomes in the children born from frozen oocytes. The research continues to look at different methods of oocyte cryopreservation. Many smaller studies have been conducted with some success but larger clinical trials are needed to replicate these findings. The conventional cryopreservation technique has been slow cooling with differing methods of freezing; however, vitrification is now being researched as the potential cryopreserving method that holds some promise for the future.

Our hypothesis is the use of vitrification (quick freezing) to cryopreserve oocytes in patients undergoing in-vitro fertilization will be more successful than slow freezing in oocyte survival, fertilization rate with ICSI and subsequent embryo development, implantation rate and pregnancy rate.

DETAILED DESCRIPTION:
Cryopreservation of oocytes is desirable because it: 1) would allow infertility patients to store excess oocytes instead of embryos, eliminating some of the ethical and religious concerns that accompany embryo storage; 2) permit storage of donor oocytes to avoid donor-recipient synchronization difficulties; and 3) can help women who may face sterilization due to chemotherapy or radiation. Oocyte cryopreservation is therefore gaining in popularity as an option for infertility treatment as well as fertility preservation.

Oocyte cryopreservation using conventional slow-cooling methods has not had much success; however more recent results have provided more optimism (Boldt et al., 2003; Porcu et al., 1997; 2000; 2002; Yang et al., 1998; 1999; 2002; Winslow et al., 2001). Vitrification has also been employed (Hong et al., 1999; Kuleshova et al., 1999; Yoon et al., 2000, 2003; Chung et al 2000; Wu et al., 2001: Kuwayama et al., 2005) with increased oocyte survival rate and live births. Vitrification is performed by suspending the oocytes in a solution containing a high concentration of cryoprotectants and then plunging them directly into liquid nitrogen (Rall and Fahy, 1985). The advantage of this technique is to prevent the formation of ice crystals within the oocyte. However the toxic effect of the high concentration of the cryoprotectant media has been a concern. New vitrification techniques which attempt to accelerate the cooling rate by decreasing the cryosolution volume and concentration, may reduce the potential toxicity. In addition, a more rapid cooling rate results in reduced chilling injury (Vajta et al., 1998).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≤ 36 years old
* Day #3 follicle stimulation hormone (FSH) < 10mIU/ml, and Estradiol < 70 pg/ml.
* The study will be limited to couples who do not wish to cryopreserve excess embryos, who would otherwise have their excess oocytes discarded.
* Body Mass Index (BMI) ≤ 35
* Patients currently being seen in our offices

Exclusion Criteria:

* Male partner requiring microsurgical epididymal sperm aspiration or testicular sperm extraction (MESA/TESE) for sperm retrieval
* Day #3 follicle stimulation hormone (FSH) > 10mIU/ml, or estradiol > 70 pg/ml
* Diagnosis of Polycystic Ovary Syndrome (PCOS)
* Body Mass Index (BMI) >35

Ages: 21 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The Center for Advanced Reproductive Services patient population
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2006-07; Primary Completion 2009-10 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Oocyte survival | When patient returns for thaw cycle

SECONDARY OUTCOMES:
Implantation rate | 2 weeks after transfer of thawed oocyte

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Benadiva, MD, HCLD, Principal Investigator — The Center for Advanced Reproductive Services, P.C.
Locations (1):
- The Center for Advanced Reproductive Services, Farmington, Connecticut, United States

REFERENCES:
- [Background] Boldt J, Cline D, McLaughlin D. Human oocyte cryopreservation as an adjunct to IVF-embryo transfer cycles. Hum Reprod. 2003 Jun;18(6):1250-5. doi: 10.1093/humrep/deg242. PMID 12773454
- [Background] Carroll J, Depypere H, Matthews CD. Freeze-thaw-induced changes of the zona pellucida explains decreased rates of fertilization in frozen-thawed mouse oocytes. J Reprod Fertil. 1990 Nov;90(2):547-53. doi: 10.1530/jrf.0.0900547. PMID 2250252
- [Background] Fuku E, Xia L, Downey BR. Ultrastructural changes in bovine oocytes cryopreserved by vitrification. Cryobiology. 1995 Apr;32(2):139-56. doi: 10.1006/cryo.1995.1013. PMID 7743816
- [Background] Hong SW, Chung HM, Lim JM, Ko JJ, Yoon TK, Yee B, Cha KY. Improved human oocyte development after vitrification: a comparison of thawing methods. Fertil Steril. 1999 Jul;72(1):142-6. doi: 10.1016/s0015-0282(99)00199-5. PMID 10428163
- [Background] Kuleshova L, Gianaroli L, Magli C, Ferraretti A, Trounson A. Birth following vitrification of a small number of human oocytes: case report. Hum Reprod. 1999 Dec;14(12):3077-9. doi: 10.1093/humrep/14.12.3077. PMID 10601099
- [Background] Porcu E, Fabbri R, Seracchioli R, Ciotti PM, Magrini O, Flamigni C. Birth of a healthy female after intracytoplasmic sperm injection of cryopreserved human oocytes. Fertil Steril. 1997 Oct;68(4):724-6. doi: 10.1016/s0015-0282(97)00268-9. PMID 9341619
- [Background] Porcu E, Fabbri R, Damiano G, Giunchi S, Fratto R, Ciotti PM, Venturoli S, Flamigni C. Clinical experience and applications of oocyte cryopreservation. Mol Cell Endocrinol. 2000 Nov 27;169(1-2):33-7. doi: 10.1016/s0303-7207(00)00348-8. PMID 11155951
- [Background] Rall WF, Fahy GM. Ice-free cryopreservation of mouse embryos at -196 degrees C by vitrification. Nature. 1985 Feb 14-20;313(6003):573-5. doi: 10.1038/313573a0. PMID 3969158
- [Background] Stachecki JJ, Cohen J, Willadsen S. Detrimental effects of sodium during mouse oocyte cryopreservation. Biol Reprod. 1998 Aug;59(2):395-400. doi: 10.1095/biolreprod59.2.395. PMID 9687313
- [Background] Stachecki JJ, Cohen J, Willadsen SM. Cryopreservation of unfertilized mouse oocytes: the effect of replacing sodium with choline in the freezing medium. Cryobiology. 1998 Dec;37(4):346-54. doi: 10.1006/cryo.1998.2130. PMID 9917351
- [Background] Stachecki JJ, Cohen J, Schimmel T, Willadsen SM. Fetal development of mouse oocytes and zygotes cryopreserved in a nonconventional freezing medium. Cryobiology. 2002 Feb;44(1):5-13. doi: 10.1016/S0011-2240(02)00007-X. PMID 12061843